CLINICAL TRIAL: NCT03700723
Title: Multicenter, Single-Blinded, Randomized, Comparator-Controlled Noninferiority Trial to Compare the Efficacy & Safety of Resusix With FP24 in Patients With Acquired Coagulopathy
Brief Title: Comparison of the Efficacy & Safety of Resusix With FP24 in Patients With Acquired Coagulopathy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Convenience of Government Funding Sponsor
Sponsor: Entegrion, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RSX-201
Record Dates: First submitted 2018-09-18; First posted 2018-10-09 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Coagulopathy
MeSH Terms: conditions — Hemostatic Disorders

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized in a 1:1 ratio to receive Resusix or FP24
Who Masked: Participant, Outcomes Assessor
Masking Description: Single blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Resusix (Experimental): The experimental drug (Resusix) will be administered intravenously to subjects enrolled in this arm of the study. Subjects may receive doses of 1-4 units during the blinded intervention period.
  Interventions: Biological: Resusix
- FP24 (Frozen Plasma) (Active Comparator): The active comparator FP24 will be administered intravenously to subjects enrolled in this arm of the study. Subjects may receive doses of 1-4 units during the blinded intervention period.
  Interventions: Biological: FP24 (Frozen Plasma)

INTERVENTIONS:
Biological: Resusix — spray-dried solvent/detergent treated plasma (blood product)
  Arms: Resusix
Biological: FP24 (Frozen Plasma) — plasma frozen within 24 hours of phlebotomy
  Arms: FP24 (Frozen Plasma)

SUMMARY:
Phase 2a study to assess the safety and efficacy of IV infused spray-dried solvent/detergent -treated plasma (Resusix) when compared with an equal volume of plasma frozen within 24 hours after phlebotomy (FP24) in patients with liver disease who are actively bleeding or who require prophylaxis for surgical bleeding

ELIGIBILITY:
Inclusion Criteria:

* SBP 90-150 mm Hg
* acquired coagulopathy due to hepatic disease
* INR >1.4
* Order for 1-4 units of plasma for active bleeding or prophylaxis for bleeding prior to surgery or invasive procedure
* Written informed consent
* MELD score: 25 or less (1st cohort), 35 or less (2nd cohort)

Exclusion Criteria:

* Pregnant women
* Incarcerated patients
* Life expectancy less than 72 hours
* Severe bleeding at time of enrollment
* HIV, sepsis, intracranial bleeding, congenital disorder, anti-phospholipid antibody syndrome or known lupus anticoagulant antibodies
* Receipt of plasma products, coagulation factor concentrates or anti-platelets within 3 days of enrollment
* Specific factor inhibitor activity or history of hypersensitivity to plasma-derived products
* Receipt of iv heparin within 24 hours of enrollment
* Use of a continuous infusion of an intravenous vasoactive medication
* Thrombocytopenia
* BMI greater than or equal to 40 kg/m2
* Participation in another clinical trial within 30 days of enrollment and received investigational product that may impact safety or efficacy of this study
* West Haven Hepatic Encephalopathy Grade 3 or 4 (cohort 1) and Grade 4 (cohort 2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-12-14 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-04-15 (Actual)

PRIMARY OUTCOMES:
Change in INR | 120 minutes
  Measured as a ratio
Total incidence of all related SAEs | 7 days
  Count of events

SECONDARY OUTCOMES:
Change in activated partial thromboplastin time (aPTT) | 72 hours
  Measured in seconds
Change in platelet count | 72 hours
  Measured in x10.e3/uL
Change in hemoglobin | 72 hours
  Measured in g/L
Change in clotting function | 72 hours
  Measured by thromboelastography (TEG) or rotational thromboelastometry (ROTEM)
Volume of plasma to correct INR | 72 hours
  Measured in mL
Time to INR reduction below 1.5 | 72 hours
  Measured in minutes
Volume of fluid (e.g., crystalloid, colloid, blood component) administered | 72 hours
  Measured in mL
Change in bleeding score in patients with active bleeding | 120 minutes
  Measured as excellent, good or poor
Thrombin generation | 72 hours
  Measured in nM
Serology for human immunodeficiency virus | 95 days
  Measured in IU/mL
Serology for hepatitis | 95 days
  Measured in IU/mL
Change in Sequential Organ Failure Assessment Score (SOFA) | 96 hours
  Measured as 0 to 4

CONTACTS AND LOCATIONS:
Overall Officials: Michael Galiger, Study Director — Entegrion, Inc.
Locations (3):
- United States (3):
  - University of Arizona, Tucson, Arizona
  - Washington University St. Louis, St Louis, Missouri
  - Carolinas Medical Center, Charlotte, North Carolina